CLINICAL TRIAL: NCT01197391
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending, Single-Dose Study of the Safety, Tolerability and Bioeffect of Subcutaneous REGN 728 in Healthy Volunteers
Brief Title: Ascending Dose Study of the Safety and Tolerability of REGN728 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R728-CL-0915
Record Dates: First submitted 2010-08-11; First posted 2010-09-09 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Dose 1 versus placebo
  Interventions: Biological: REGN728
- Cohort 2 (Experimental): Dose 2 versus placebo
  Interventions: Biological: REGN728

INTERVENTIONS:
Biological: REGN728 — 2 Subcutaneous Cohorts (dose 1, 2)

SUMMARY:
This study will test the safety and tolerability (how the body reacts to the drug) of REGN728 compared with placebo (an inactive substance that contains no medicine) in healthy subjects. The study drug and placebo will be administered by subcutaneous injection (under the skin) at the clinic visit. There will be 14 clinic visits, which will include 4 overnight stays. Subjects will be monitored by the study staff for side effects and the body's response to the study drug. Vital signs (blood pressure, temperature, breathing and heart rate) will be checked, blood and urine samples will be collected at some or all visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 65 years of age.
* Weight> 50 kg and <95 kg inclusive
* For men of childbearing potential, willingness to utilize adequate contraception and not have their partner[s] become pregnant during the full duration of the study.
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
* Able to read, understand and willing to sign the informed consent form.

Exclusion Criteria:

* Initiation of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to screening visit.
* Women of childbearing potential, pregnant and breast-feeding women are excluded. Women are considered to be of childbearing potential until they have been amenorrheic for at least 12 months or have had surgical sterilization.
* Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that would adversely affect the subject's participation in this study.
* Hospitalization for any reason within 60 days of screening.
* Known history of Human Immunodeficiency Virus (HIV) antibody; and/or positive Hepatitis B surface antigen, and/or positive Hepatitis C antibody at the screening visit.
* Previous exposure to any therapeutic or investigational biological agent.
* History of alcohol or substance abuse within a year prior to the screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study is the percentage of subjects with treatment emergent adverse events, reported from the administration of study drug on day 1 to the completion of the study on day 106. | 106 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Miramar, Florida
  - Overland Park, Kansas